CLINICAL TRIAL: NCT00870649
Title: Efficacy and Safety Evaluation of the Therapeutic Vaccine Candidate Sh28GST in Association With Praziquantel (PZQ) for Prevention of Clinical and Parasitological Recurrences of S. Haematobium Infection in Children
Brief Title: Efficacy of Bilhvax in Association With Praziquantel for Prevention of Clinical Recurrences of Schistosoma Haematobium
Acronym: Bilhvax3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BT05-01; 2008-006757-40 (EudraCT Number)
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2016-11

CONDITIONS: Urinary Schistosomiasis; Schistosoma Haematobium
Keywords: Schistosomiasis vaccine; therapeutic vaccine; Bilhvax
MeSH Terms: conditions — Schistosomiasis haematobia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bilhvax vaccine (Sh28GST) (Experimental): Arm 1 : S. haematobium infected children pretreated by two doses of PZQ (at Week-9 and W-8)receiving 3 injections of candidate vaccine at D0, W4, W8 and a boost at W52, and then treated by a third dose of PZQ at W44.
  Interventions: Biological: Bilhvax vaccine (Sh28GST)
- Placebo (Placebo Comparator): Arm 2 : S. haematobium infected children pretreated by two doses of PZQ (at Week-9 and W-8)receiving 3 injections of placebo at D0, W4, W8 and a boost at W52, and then treated by a third dose of PZQ at W44.
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: Bilhvax vaccine (Sh28GST) — Four vaccine sc administrations over a year associated with chemotherapy (PZQ)
  Arms: Bilhvax vaccine (Sh28GST)
Biological: placebo — Four placebo sc administrations over a year associated with chemotherapy (PZQ)
  Arms: Placebo

SUMMARY:
Objectives:To reduce the risk of S. haematobium pathology recurrences during the three years following vaccine administration and to control the safety of this therapeutic strategy in children exposed to urinary schistosomiasis.

Methodology : Phase III trial, self-contained, randomized, double blind, in two parallel groups receiving 3 injections at D0, W4, W8 and a boost at W52, one group receiving "Bilhvax", the other one placebo, in S. haematobium infected children pretreated by two doses of PZQ (at W9 and W8) Patient included : Infected school children, 6 to 9 years of age.

Primary objective : To demonstrate a significant delay of recurrence of the schistosomiasis pathology in vaccine group compared to control group in the 3 years period following the first administration (between D0 and W152).

Secondary objective : safety

Duration : February 2009 to March 2012

DETAILED DESCRIPTION:
Patient inclusion (detailed criteria):

Children in CI or CP classes of public schools in St Louis Region (Senegal) A male or female between, and including, 6 and 9 years of age at the time of the first vaccination Free of obvious health problems excepted schistosomiasis as established by clinical examination (W8-W1) Found positive for S. haematobium infection during the selection period (W12 à W9) : microhaematuria ≥ 2+ et Urinary Filtration, UF ≥ 50 eggs of Sh/10ml urine Written inform consent obtained from the parent or guardian of the subject (W9) and child acceptance Pretreated with 2 doses of 40mg/kg PZQ (at W9 and W8) Absence of heavy lesions of the urinary tract under echotomography (W8 et W1)

Primary objective (detailed):

To demonstrate a significant delay of recurrence of the schistosomiasis pathology in vaccine group compared to control group in the 3 years period following the first administration (between D0 and W152).

Criterion of meeting the recurrence is the association of :

Positive microscopic haematuria (positivity by urinary stick : ≥ 1+)

* either during the active visits (W82, W100, W117, W134, or W152).
* or after spontaneous complaint of the patient at any time Positive parasitological test defined as the presence of at least one living egg of S. haematobium during one out of three UF (one UF per day/3 days during one week). The delay of the first recurrence is defined as the delay between the date of inclusion and the date of the positive parasitological test.

Statistical considerations : The number of patients necessary to detect the expected difference after 3 years of study (50% of recurrence in vaccinated group versus 70% in placebo group), with a statistical power of 80% and a bilateral test at 5%, is 103 children per group. To assume the lost of statistical power in the "intention to treat" analysis (ITT) resulting from the number of cases where vaccine protocol has not been completed, 125 children per group will be included in the study. In total 250 children will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Children in CI or CP classes of public schools in St Louis Region (Senegal) A male or female between, and including, 6 and 9 years of age at the time of the first vaccination Free of obvious health problems excepted schistosomiasis as established by clinical examination (W8-W1) Found positive for S. haematobium infection during the selection period (W12 à W9) : microhaematuria ≥ 2+ et Urinary Filtration, UF ≥ 50 eggs of Sh/10ml urine Written inform consent obtained from the parent or guardian of the subject (W9) and child acceptance Pretreated with 2 doses of 40mg/kg PZQ (at W9 and W8) Absence of heavy lesions of the urinary tract under echotomography (W8 et W1)

Exclusion Criteria:

* Absence of written inform consent or expressed refusal from the child Vaccination other than the study vaccine within 90 days preceding the first dose of study vaccine, or planned use during the study period.

Chronic administration (defined as more than 14 days) of immunosuppressants or other immuno-modifying drugs, actual or since previous year.

History of allergic disease or reactions likely exacerbated by any component of the vaccine Acute disease at time of enrolment Other conditions which in opinion of the PI may potentially represent a danger for the child to be enrolled.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Actual)
Dates: Start 2009-02; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
A significant delay of recurrence of the schistosomiasis pathology in vaccine group compared to control group. | Evaluation three years after first administration

SECONDARY OUTCOMES:
Evaluation of safety Percentage of children presenting at least one adverse event of degree ≥ 2. Percentage of children presenting at least one adverse event implying modification of the vaccine strategy. | During the three year study

CONTACTS AND LOCATIONS:
Overall Officials: Gilles RIVEAU, PhD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- ESPOIR Pour La Santé, Saint-Louis, Senegal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Riveau G, Schacht AM, Dompnier JP, Deplanque D, Seck M, Waucquier N, Senghor S, Delcroix-Genete D, Hermann E, Idris-Khodja N, Levy-Marchal C, Capron M, Capron A. Safety and efficacy of the rSh28GST urinary schistosomiasis vaccine: A phase 3 randomized, controlled trial in Senegalese children. PLoS Negl Trop Dis. 2018 Dec 7;12(12):e0006968. doi: 10.1371/journal.pntd.0006968. eCollection 2018 Dec. PMID 30532268